CLINICAL TRIAL: NCT00813839
Title: Comparison of Automated Ventilator Controlled Weaning to Daily Spontaneous Breathing Trial Weaning Protocol in ICU Patients Following Prolonged Mechanical Ventilation.
Brief Title: Automated Ventilator Controlled Weaning vs Daily Spontaneous Breathing Trial in Difficult to Wean ICU Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: for inability to enroll subjects.
Sponsor: University of California, San Francisco (Other)
Responsible Party: Jenson Wong MD, Department of Anesthesia, UCSF
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H60971-32402-02
Record Dates: First submitted 2008-12-19; First posted 2008-12-23 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Mechanical Ventilation; Weaning
Keywords: SmartCare; Spontaneous Breathing Trials; Mechanical Ventilation; Weaning; Patients requiring prolonged mechanical ventilation (>72 hours)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 SmartCare (Experimental): automated ventilator controlled adjustment of pressure support
  Interventions: Other: daily weaning trails
- 2 spontaneous breathing Trial (Active Comparator): daily SBT on minimum pressure support
  Interventions: Other: daily weaning trails

INTERVENTIONS:
Other: daily weaning trails — daily SmartCare vs SBT until extubation criteria met

SUMMARY:
This study will compare Drager Smart Care (SC), a commercially available automated ventilator controlled weaning mode to the current daily spontaneous breathing trial (SBT) weaning protocol. The study is designed to determine if automated ventilator controlled weaning can reduce total duration of intubation following mechanical ventilation in ICU patients requiring prolonged mechanical ventilation (>72 hours).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Intubated with endotracheal tube
* Requiring mechanical ventilation for > 72 hours
* Meets weaning criteria: Improvement or resolution of the underlying process that precipitated need for mechanical ventilation, PaO2 ≥ 60 mm Hg on PEEP and FiO2 Requirements of ≤ 8 cm H2O and FiO2 ≤ 0.50, Stable oxygenation: PEEP and FiO2 requirements not increased in the past 24 hrs, Ability to initiate an inspiratory effort and trigger the ventilator, Subject enrollment approved by the primary service attending physician

Exclusion Criteria:

* Pregnancy
* Patients with tracheostomy or planned tracheostomy prior to attempt to extubate
* Patients with known airway patency issues that are anticipated to delay extubation.
* Patients with neurological injury in whom care is likely to be withdrawn
* Patients with cervical spinal cord injury.
* Prospective subject or surrogate consenter does not fully understand the implications of the study because of a language barrier.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-11; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
weaning time to successful spontaneous breathing trial | 28 days or extubation
weaning time to successful extubation | 28 days or extubation
ventilator weaning days | 28 days or extubation
total duration of ventilatory support | 28 days or extubation

SECONDARY OUTCOMES:
reintubations within 48 hours | 48 hrs
sedation and analgesic requirements | 28 days or extubation
ICU and hospital length of stay | total time of ICU and hospital stay
clinical staff time requirements | during active weaning period

CONTACTS AND LOCATIONS:
Locations (1):
- San Francisco General Hospital, UCSF Dept. of Anesthesia, San Francisco, California, United States